CLINICAL TRIAL: NCT02676739
Title: A Double-blind Placebo Controlled Study of Mixed-amphetamine Salts, Extended Release (Adderall XR) for Cognitive Impairment in MS
Brief Title: Adderall XR and Cognitive Impairment in MS
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sarah Morrow (Other)
Responsible Party: Sponsor-Investigator, Sarah Morrow, Principal Investigator, London Health Sciences Centre
Organization: London Health Sciences Centre (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10012443
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — SLI381

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Capsule with no active medical ingredients to be taken orally once a day for 12 weeks.
  Interventions: Drug: Adderall XR
- Adderall XR 10mg (Active Comparator): 10mg Adderall XR capsule to be taken orally once a day for 12 weeks.
  Interventions: Drug: Adderall XR
- Adderall XR 20mg (Active Comparator): 20mg Adderall XR capsule to be taken orally once a day for 12 weeks.
  Interventions: Drug: Adderall XR

INTERVENTIONS:
Drug: Adderall XR

SUMMARY:
This 12 week randomized placebo-controlled study will compare the effects of 10 mg and 20 mg of a mixed amphetamine salt, extended release medication (trade name Adderall XR) to placebo on objective measures of processing speed and memory, as well as on self-reported measures of cognition and quality of life. To be enrolled in the study, MS subjects must demonstrate impaired processing speed on the Symbol Digit Modalities Test (SDMT).

DETAILED DESCRIPTION:
It is now known that Multiple Sclerosis (MS) can cause cognitive impairment (CI), estimated to occur in 40-65% of MS patients. The most frequently observed impairments in the MS population are in processing speed (PS), as well memory (working and episodic), verbal fluency, executive function and selective attention can also be involved. Longitudinal studies demonstrate a slowly progressive, insidious course; thus CI is unlikely to remit once present. CI has a negative effect on personal relationships and self-esteem, leading to social isolation. Also, a decrease in PS over time predicts a decrease in employment status in MS patients. Thus, CI is an important, but under-recognized consequence of MS and yet there are currently no approved therapies to treat this common symptom.

Amphetamines represent a candidate class of drugs to treat CI in patients with MS, based on both animal and human studies. Amphetamines are the standard of care for attentional/PS deficits in attention deficit (hyperactivity) disorder (ADHD) and multiple studies demonstrate an increase in speed and accuracy, as well as performance on daily activities. Previous studies in the MS population have demonstrated mixed results, which may be due to different formulations of the stimulant drug. This study's lead PI recently completed a pre-post dose study with a mixed amphetamine salts formulation with an extended release delivery system (MAS-XR), trade name Adderall XR, in an MS population with impaired PS, comparing improvement on the Symbol Digit Modalities Test (SDMT) as a result of a single dose of MAS-XR (5 mg or 10 mg) or placebo. We found that 10 mg MAS-XR significantly improved performance on the SDMT, a reliable measure of PS in the MS population. MAS-XR 10 mg resulted in an increase on the SDMT of 5.2 (± 4.5) points compared to only 0.6 (± 4.4) points in the placebo group (p = 0.047), resulting in an effect size of 0.47. However, this pilot study, due to the single dose administration, was unable to determine if this benefit is maintained over time, or examine if there is an increase in the subjective impression of change or has an effect on daily living. Thus, although promising, this previous pilot study with MAS-XR was unable to determine if the increase noted on the SDMT, an objective measure of PS, translates into any clinically meaningful impact for the person with MS.

The goal of this study is to evaluate the efficacy and safety of 10 mg and 20 mg MAS-XR for PS and memory measures in MS patients in a multi-center, randomized, placebo-controlled trial over a 12 week period across 5 sites in Canada. MAS-XR is composed of amphetamine sulfate salts in a 3:1 ratio of d to l-isomers of amphetamine, with time to reach maximum plasma concentration (Tmax) of 7 hours. This study, in addition to objective measures of cognitive function, will also evaluate quality of life (QoL) and subjective measures of cognitive function. We propose to recruit 180 subjects to this study, based on the sample size calculation and a potential 15% drop out, resulting in approximately 150 subjects completing the full study. Subjects will be recruited from the London (ON) MS clinic and MS cognitive clinic, lead site; Sunnybrook MS clinic (Toronto, ON); Edmonton (AB) MS clinic; Calgary (AB) MS clinic and the Dalhousie (Halifax, NS) MS clinic. Block randomization will be used. Subjects with MS of any type demonstrating impaired PS on the SDMT, who have no other medical condition that could explain this impairment, are eligible for participation. Major depression, uncontrolled or labile hypertension, a history of heart disease, or a diagnosis of bipolar disorder will result in exclusion. Daily opioid use, benzodiazepine use, other than at night, or frequent marijuana use will also result in exclusion. The primary outcome will be the SDMT, which will be measured at baseline, as well as six and 12 weeks later. Secondary outcomes will include both objective and subjective measures. The objective cognitive measures for memory will be the Brief Visuospatial Memory Test Revised (BVMTR) and California Verbal Learning Test 2nd edition (CVLT2), immediate recall (IR) measures only. The subjective measures will be the Multiple Sclerosis Neuropsychological Screening Questionnaire (MSNQ), the Perceived Deficits Questionnaire (PDQ), the 36-Item Short Form Survey (SF-36), the Modified Fatigue Impact Scale (MFIS) and the Hospital Anxiety and Depression Scale (HADS) as measures of different aspects of QoL, administered at baseline and 12 weeks later. Adverse events, as well as heart rate and blood pressure, will be investigated at each study visit.

Overall, this study addresses a significant consequence of MS, cognitive impairment, a symptom that can have a devastating impact on quality of life and the ability of MS patients to fully participate in their community. Once present, CI is unlikely to remit, likely to progress, and currently has no proven treatment. The previous pilot study conducted by the lead PI with MAS-XR demonstrates that it is a promising potential treatment for processing speed impairment in MS patients. This study builds on the previous pilot data, improving the ability to determine if MAS-XR is a safe and effective treatment for CI for the MS population.

ELIGIBILITY:
Inclusion Criteria:

* MS of any type as per 2010 McDonald's criteria
* Males/females between the ages of 18-59, inclusive
* Have not received corticosteroids or experienced a relapse in the last ninety days
* An Expanded Disability Status Scale (EDSS) of ≤ 7.0
* If female, must neither be pregnant nor breast-feeding (pregnancy test to be complete at enrollment for those of childbearing potential)
* Willingness to use appropriate contraceptive measures (hormonal contraceptives (i.e., oral contraceptives, patch, vaginal ring, injectables or implants); intrauterine device or system; vasectomy or tubal ligation) both males and females at least 28 days before, for the duration of the trial and for at least 30 days after the study ends unless post-menopausal (no menses for 12 months) or surgically sterile female (complete hysterectomy, bilateral salpingectomy, or tubal ligation with documentation) or vasectomised male partner (with appropriate documentation of azoospermia).
* Ability to complete the neuropsychological tests included in the battery including binocular visual acuity of ≤ 20/70 corrected or uncorrected
* Stable medications for over the last 30 days with no planned change for the duration of the study.

Exclusion Criteria:

* Evidence of other medical potential cause(s) of cognitive deficits such ADHD, TBI, Alzheimer's disease or other dementia, stroke, previous chronic CNS infection or other neurological disorders
* Evidence of untreated major depression as by clinician interview or patient report
* Family history of suicide, major depression, or bipolar disorder
* Uncontrolled or labile hypertension (> 135/85 mmHg), treated or untreated
* History of structural heart disease, including atherosclerosis or angina
* Diagnosis of bipolar disorder or a history of a psychotic episode
* Daily opioid use
* Daily benzodiazepine use other than nightly administration
* Use of other amphetamine or other sympathomimetic medication
* Use of naturally grown medicinal or non-medicinal marijuana more than 3x/week or 14x/month
* those with Hyperthyroidism or Glaucoma
* A history of drug abuse
* Known hypersensitivity to sympathomimetic amines
* A history of agitated or aggressive states
* Those taking monoamine oxidase inhibitors or other drugs that may interact with the study medication
* A known allergy to amphetamines or components of Adderall XR or container
* Past or present suicidal behavior or ideation
* Those with renal impairment or on nephrotoxic drugs.
* Have motion tics (hard to control, repeat twitching of any parts of the body) or verbal tics (hard to control repeating of sounds or words) or Tourette's syndrome
* Family history motion tics, verbal tics, or Tourette's syndrome
* Family history of sudden death, QT prolongation
* Positive pregnancy test
* Beck Depression Inventory - Fast Screen score question 7 marked 2 or 3 by participant, or scores in the severe range

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-05-20 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Symbol Digit Modalities Test (SDMT) | 12 weeks
  This task will be performed at enrollment (and baseline if enrollment occurred great than 7 days prior), week 6 and week 12 after starting the medication. The SDMT is one of the most commonly used tests to assess processing speed in the MS population and is included in the two validated neuropsychological test batteries routinely used in MS studies, the Minimal Assessment of Cognitive Function in MS (MACFIMS).

SECONDARY OUTCOMES:
Brief Visuospatial Memory Test Revised - immediate recall | 12 weeks
  A measure of visual/spatial memory with 3 recall trials of the same six figures, marked for accuracy of the figure drawn and their spatial location on the page. Assessed at baseline and after taking the study medication for 12 weeks.
California Verbal Learning Test 2nd edition - immediate recall | 12 weeks
  Assesses auditory/verbal memory, with five learning trials of the same 16 words. It is scored as the total number of words recalled, or learned, for each of the 5 trials. Assessed at baseline and after taking the study medication for 12 weeks.
Multiple Sclerosis Neuropsychological Screening Questionnaire | 12 weeks
  Is a 15 item self-report questionnaire designed to screen for cognitive impairment (CI) in MS subjects. The questions all relate to cognitive problems in daily life and are scored from 0 (never, does not occur) to 4 (very often, very disruptive) and a composite score is calculated, thus higher numbers indicate greater perceived CI. Assessed at baseline and after taking the study medication for 12 weeks.
Perceived Deficits Questionnaire | 12 weeks
  developed specifically for the MS population to cover the domains of cognitive function most often impaired in MS: attention, retrospective and prospective memory, as well as planning and organization. It is a 20 item self-report questionnaire that is scored from 0 (never occurs) to 4 (almost always). Assessed at baseline and after taking the study medication for 12 weeks.
36-Item Short Form Survey | 12 weeks
  Considered as the gold standard generic measure of health status, and has been used extensively in MS Quality of Life (QoL) research. This self-report questionnaire provides 2 summary scores: physical and mental component summary scores, with higher scores indicating better perceived health-related quality of life. It has been used to detect effects of treatment in different patient populations and discriminates between levels of disease severity. Assessed at baseline and after taking the study medication for 12 weeks.
The Modified Fatigue Impact Scale | 12 weeks
  A measure of fatigue assessed at baseline and 12 weeks after the study medication. It is a 21 item questionnaire that assesses the perceived impact of fatigue on activities of daily life, and can be reported as a total score or divided into 3 subscales (physical, cognitive and psychosocial), with higher scores indicating higher levels of fatigue. Fatigue is less likely to affect objective cognitive assessments, but there is some evidence that it can affect performance on the SDMT
Hospital Anxiety and Depression Scale | 12 weeks
  A measure of anxiety and depression, assessed at baseline and 12 weeks after taking the study medication. There are 14 questions in total, scoring responses from 0-3 reflecting the severity of the symptom. The two sub-scores, HADS-A (anxiety) and HADS-D (depression) both ranging from 0-21, have been validated in the MS population. Depression is well known to impact cognitive function, including in the domains included in the study; less has been studied regarding the impact of anxiety but recent cross-sectional studies suggest the presence of anxiety is correlated with lower performance on objective cognitive tests.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

REFERENCES:
- [Background] Morrow SA, Rosehart H. Effects of single dose mixed amphetamine salts--extended release on processing speed in multiple sclerosis: a double blind placebo controlled study. Psychopharmacology (Berl). 2015 Dec;232(23):4253-9. doi: 10.1007/s00213-015-4051-6. Epub 2015 Aug 21. PMID 26289355